CLINICAL TRIAL: NCT01644292
Title: Enhancing Participation In the Community by Improving Wheelchair Skills (EPIC WheelS): Phase 2
Brief Title: Enhancing Participation In the Community by Improving Wheelchair Skills: Phase 2
Acronym: EPIC WheelS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2012:069
Record Dates: First submitted 2012-07-13; First posted 2012-07-19 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2014-01

CONDITIONS: Older Adult Manual Wheelchair Users
Keywords: Mobility Impairment; Manual Wheelchair; Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPIC Wheels Training Intervention (Experimental): EPIC Wheels skills training program
  Interventions: Other: EPIC WheelS

INTERVENTIONS:
Other: EPIC WheelS — EPIC WheelS is a user-centred program for wheelchair skills training that combines two structured 1-hour sessions with an expert trainer and four weeks of self-directed practice and training in the natural (home) environment.

SUMMARY:
The purpose of this project is to conduct a pilot study of the EPIC WheelS wheelchair skills home training program for older adults in preparation for a third phase feasibility study.

DETAILED DESCRIPTION:
Many older adults rely on a manual wheelchair for community mobility but are not provided with skills for independent and effective use. Suboptimal or disuse of the wheelchair results in substantial social costs such as reduced engagement in meaningful activity, social isolation, and higher caregiver burden. This represents a poor use of financial resources, including the cost of wheelchair acquisition and demands for attendant care. Access to skills training is constrained by the cost and limited availability of skilled therapists, the demands of patient and clinician travel, and lack of programs designed specifically for the needs of older adults. Enhancing Participation In the Community by improving Wheelchair Skills (EPIC WheelS) is an individualized home-training program that optimizes learning for older adults while limiting the demands on expert clinician trainers. It is delivered using a portable computer tablet that allows interactive learning, customized updating, and communication with an expert trainer. A monitored, home program that is effective and efficient for older adults has potential application for other target groups as well, particularly those with limited access to rehabilitation services in rural and remote locations.

ELIGIBILITY:
Inclusion Criteria:

* at least 50 years old
* live in the community within metropolitan Winnipeg
* self-propel a MWC (Manual Wheelchair) at least 1 hour per day
* use their MWC for mobility outside of the home
* have used a MWC for less than 2 years

Exclusion Criteria:

* cannot communicate and complete study questionnaires in English
* anticipate a health condition that contraindicates wheelchair training

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed M Giesbrecht, PhD (Cand.), Principal Investigator — University of Manitoba; William C Miller, PhD, Principal Investigator — University of British Columbia; Janice Eng, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Giesbrecht EM, Miller WC, Jin BT, Mitchell IM, Eng JJ. Rehab on Wheels: A Pilot Study of Tablet-Based Wheelchair Training for Older Adults. JMIR Rehabil Assist Technol. 2015 Apr 30;2(1):e3. doi: 10.2196/rehab.4274. PMID 28582240

RESULTS

PARTICIPANT FLOW:
Groups:
- Training Intervention: EPIC WheelS : EPIC WheelS is a user-centred program for wheelchair skills training that combines two structured 1-hour sessions with an expert trainer and four weeks of self-directed practice and training in the natural (home) environment.
Period: Overall Study
Arm/Group | Training Intervention
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Training Intervention
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Wheelchair Skills Test (WST) 4.1 Capacity Score
Description: The WST is a structured assessment with 32 discrete mobility skills required to perform social roles in the community, each scored dichotomously as pass/fail. The WST produces a total Skill Capacity score (0-100%) reflecting the number of skills safely passed.
Time Frame: Baseline and follow-up (1 month)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 2
units on a scale | 6.25 (8.84)

ADVERSE EVENTS:
Arm/Group | Training Intervention
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes